CLINICAL TRIAL: NCT02804724
Title: Factors Associated With Late HIV Diagnosis in Grampian: an Epidemiological Study
Status: Completed | Type: Observational
Sponsor: University of Aberdeen (Other)
Collaborators: NHS Grampian (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2-030-15
Record Dates: First submitted 2015-06-29; First posted 2016-06-17 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-06

CONDITIONS: Human Immunodeficiency Virus
Keywords: HIV; Human immunodeficiency virus; Late diagnosis
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Newly diagnosed individuals with HIV: Individuals newly diagnosed with HIV in Grampian between January 2009 and December 2014
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
Human immunodeficiency virus (HIV) is a major global health concern which has resulted in an estimated 39 million deaths world-wide. Although it is now a treatable medical condition there is still avoidable morbidity and mortality associated with HIV infection in the UK. Late diagnosis (CD4 count of <350 cells/mm3 or AIDS-defining illness irrespective of CD4 count) is associated with increased morbidity and mortality, increased risk of transmission, impaired response to antiretroviral therapy and increased healthcare costs. In Grampian, 49% of patients were diagnosed late between 1984 and 2011. Therefore, the aim of the study is to determine the factors associated with late HIV diagnosis in Grampian between 2009 and 2014 to ascertain whether diagnoses could have been made earlier.

The study constitutes a secondary data analysis. Individuals newly diagnosed with HIV between January 2009 and December 2014 were identified from a Health Protection Scotland (HPS) database. The majority of outcome data were extracted from the existing HPS database. Missing data were collected via a retrospective review of patient case-notes, laboratory reports and an electronic patient management system. Patients were classified as early or late diagnosis and comparisons were made between the groups using statistical tests. The study sought to provide a basis for recommendations for improvement of information and services to facilitate earlier HIV diagnosis in Grampian.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with HIV between January 2009 and December 2014
* Individuals diagnosed in NHS Grampian

Exclusion Criteria:

* Individuals aged < 16 years of age

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals newly diagnosed with HIV in Grampian between January 2009 and December 2014
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2015-06; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Age at diagnosis | 5 years
  Age in years at diagnosis; compared between early and late diagnosis groups.
Gender | 5 years
  Gender; compared between early and late diagnosis groups
Scottish Index of Multiple Deprivation (SIMD) Quintile | 5 years
  SIMD quintile (1 representing most deprived to 5 representing least deprived); compared between early and late diagnosis groups
Ethnicity | 5 years
  Ethnic group; compared between early and late diagnosis groups
Migrant status | 5 years
  Migrant status in relation to the United Kingdom; compared between early and late diagnosis groups
Probable mode of transmission | 5 years
  Probable mode of HIV transmission; compared between early and late diagnosis groups
Probable region of exposure | 5 years
  Probable region of exposure to HIV; compared between early and late diagnosis groups
Registration with General Practitioner | 5 years
  Current registration status with General Practitioner; compared between early and late diagnosis groups
Contact with healthcare professional | 5 years
  Contact with healthcare professional(s) in the year preceding HIV diagnosis (contact versus no contact); compared between early and late diagnosis groups
Frequency of healthcare contacts | 5 years
  Frequency of contact with healthcare professional(s) in the year preceding HIV diagnosis; compared between early and late diagnosis groups
Previous HIV testing | 5 years
  Previous HIV testing (no testing versus testing); compared between early and late diagnosis groups
Clinical indicator disease | 5 years
  Presence or absence of a BHIVA clinical indicator disease in the five years preceding diagnosis; compared between early and late diagnosis groups
Number of clinical indicator disease(s) | 5 years
  Number of BHIVA clinical indicator disease(s) present in the five years preceding diagnosis; compared between early and late diagnosis groups
Co-existing hepatitis B/C infection | 5 years
  Presence or absence of a co-existing hepatitis B/C infection; compared between early and late diagnosis groups

SECONDARY OUTCOMES:
Frequency of missed opportunities for diagnosis | 5 years
  Number of missed opportunities for diagnosis as defined by the BHIVA testing guidelines; compared between early and late diagnosis groups
Circumstance of HIV diagnosis | 5 years
  Circumstance of HIV diagnosis; no BHIVA clinical indicator disease present versus testing offered following detection of a BHIVA clinical indicator disease versus no testing offered following the detection of a BHIVA clinical indicator disease. Compared between early and late diagnosis groups

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Okpo, MBBS FFPH, Principal Investigator — NHS Grampian and University of Aberdeen
Locations (1):
- NHS Grampian, Aberdeen, Aberdeen City, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wohlgemut J, Lawes T, Laing RB. Trends in missed presentations and late HIV diagnosis in a UK teaching hospital: a retrospective comparative cohort study. BMC Infect Dis. 2012 Mar 28;12:72. doi: 10.1186/1471-2334-12-72. PMID 22455558
- [Background] Sullivan AK, Curtis H, Sabin CA, Johnson MA. Newly diagnosed HIV infections: review in UK and Ireland. BMJ. 2005 Jun 4;330(7503):1301-2. doi: 10.1136/bmj.38398.590602.E0. Epub 2005 May 13. No abstract available. PMID 15894552
- [Background] Ellis S, Curtis H, Ong EL; British HIV Association (BHIVA); BHIVA Clinical Audit and Standards sub-committee. HIV diagnoses and missed opportunities. Results of the British HIV Association (BHIVA) National Audit 2010. Clin Med (Lond). 2012 Oct;12(5):430-4. doi: 10.7861/clinmedicine.12-5-430. PMID 23101142
- [Background] Lucas SB, Curtis H, Johnson MA. National review of deaths among HIV-infected adults. Clin Med (Lond). 2008 Jun;8(3):250-2. doi: 10.7861/clinmedicine.8-3-250. PMID 18624028